CLINICAL TRIAL: NCT02354547
Title: A Phase I Study of SGT-53, a TfRscFv-Liposome-p53 Complex, in Children With Refractory or Recurrent Solid Tumors
Brief Title: A Study of SGT-53 in Children With Refractory or Recurrent Solid Tumors
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: SynerGene Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGT53-01-2
Record Dates: First submitted 2014-12-18; First posted 2015-02-03 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Topotecan; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SGT-53 with Topotecan/Cyclophosphamide (Experimental): There will be 4-6 cycles (21 days/cycle) of therapy in this trial. In cycle 1, SGT-53 will be given as a single agent twice weekly starting at 1.4 mg/m² of DNA per infusion to evaluate single-agent toxicity. Pharmacokinetic studies will be performed. In the absence of dose limiting toxicity, patients will proceed to cycle 2 even if they have progressive disease. Starting in cycle 2, SGT-53 will be administered twice-weekly in combination with topotecan and cyclophosphamide administered daily for 5 days, days 1-5 of each cycle. Day 1 of each combination cycle is the first day on which topotecan and cyclophosphamide are administered with SGT-53. If a subject has at least stable disease after four cycles of therapy and is tolerating protocol therapy, two additional cycles may be considered.
  Interventions: Genetic: SGT-53; Drug: Topotecan; Drug: Cyclophosphamide

INTERVENTIONS:
Genetic: SGT-53 — The starting dose of SGT-53 will be 1.4 mg DNA/m² (dose level 1). If MTD is reached at dose level 1, subsequent cohort will be treated at 0.7 mg DNA/m² (dose level -1). If MTD is not reached at 2.1 mg DNA/m² (dose level 2), additional dose level(s) may be added. Intra-patient escalation is not allowed. Topotecan/cyclophosphamide will not be administered in cycle 1. In cycle 2, SGT-53 will be administered in combination with 0.6 mg/m² topotecan and 200 mg/m² cyclophosphamide IV daily for 5 days. Beginning in cycle 3, if no DLTs in cycle 2, topotecan and cyclophosphamide will be escalated to 0.75 mg/m² and 250 mg/m², respectively. No further dose escalation is permitted. If DLT develops at the higher doses, the doses should be decreased back to those in cycle 2.
Drug: Topotecan — Topotecan/cyclophosphamide will not be administered in cycle 1. In cycle 2, 0.6 mg/m² topotecan will be administered in combination with SGT-53 and cyclophosphamide IV daily for 5 days. Beginning in cycle 3, if no DLTs in cycle 2, topotecan will be escalated to 0.75 mg/m². No further dose escalation is permitted. If DLT develops at the higher doses, the dose should be decreased back to those in cycle 2.
  Other Names: Hycamtin
Drug: Cyclophosphamide — Topotecan/cyclophosphamide will not be administered in cycle 1. In cycle 2, 200 mg/m² cyclophosphamide will be administered in combination with topotecan and SGT-53 IV daily for 5 days. Beginning in cycle 3, if no DLTs in cycle 2, cyclophosphamide will be escalated to 250 mg/m². No further dose escalation is permitted. If DLT develops at the higher doses, the dose should be decreased back to those in cycle 2.
  Other Names: Cytoxan®; Neosar®

SUMMARY:
The purpose of this study is to determine the dose limiting toxicities and recommended phase 2 dose of SGT-53 alone and in combination with topotecan and cyclophosphamide in pediatric patients with recurrent or refractory solid tumors.

DETAILED DESCRIPTION:
The p53 is a vital human tumor suppressor gene. Loss of p53 suppressor function is present in the majority of human cancers. The p53 protein has a diverse range of functions including regulation of cell cycle checkpoints, cell death (apoptosis), senescence, DNA repair, maintenance of genomic integrity, and control of angiogenesis. Abnormalities of the p53 gene may impact the efficacy of standard anticancer treatments such as radiation and chemotherapy. P53 mutation and pathway dysfunction are associated with poor clinical outcomes and the presence of the p53 mutation correlates with resistance to chemotherapy and radiation. The development of somatic gene therapy has created the potential to restore wild type function of p53. SGT-53 is a complex of cationic liposome encapsulating a normal human wild type p53 DNA sequence in a plasmid backbone. This complex has been shown to efficiently and specifically deliver the p53 cDNA to the tumor cells. Introduction of the p53 cDNA sequence is expected to restore wtp53 function in the apoptotic pathway. P53 restoration has been shown most effective in enhancing cytotoxicity in combination with an agent which results in DNA damage or initiates apoptosis. Though mutated p53 is uncommon in childhood cancer, children with adrenocortical tumor and rhabdomyosarcoma have been found to have p53 mutations. Additionally, wild type p53 may be suppressed in tumors through pathway crosstalk. For example, in sarcomas, a common childhood solid tumor, activation of MDM2 effectively inactivates p53. Thus, the treatment proposed in this trial to reintroduce p53 may offer benefit even in patients with p53 wild-type tumors. Moreover, the SGT-53 treatment can significantly sensitize pediatric cancer cell lines to the killing effect of the standard chemotherapeutic agents, topotecan and cyclophosphamide. Thus, we propose to assess the efficacy of this combination therapy in pediatric patients with refractory or recurrent solid tumors. This phase I clinical trial is to determine the dose limiting toxicities (DLT), recommended phase 2 dose, and maximum tolerated dose (MTD) of SGT-53 (if reached) alone and in combination with conventional chemotherapy in pediatric patients with recurrent or refractory solid tumors. In addition, pharmacokinetics of escalating doses of SGT-53 is studied.

ELIGIBILITY:
Inclusion Criteria:

* All patients and/or their parents or legally authorized representatives must sign a written informed consent.
* Patients must be > than 12 months and ≤ 21 years of age at the time of study enrollment.
* Body surface Area (For Dose Level -1): Patients must be ≥ 0.38 m² at the time of study enrollment.
* Patients with relapsed or refractory solid tumors (excluding primary central nervous system tumors) are eligible. Patients must have had histologic verification of malignancy at original diagnosis or relapse.
* Patients must have either measurable or evaluable disease.
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life.
* Karnofsky ≥ 50% for patients > 16 years of age and Lansky ≥ 50 for patients ≤ 16 years of age.
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy:

  * At least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea).
  * At least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor.
  * At least 7 days after the last dose of a biologic agent.
  * At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines.
  * At least 3 half-lives of the antibody after the last dose of a monoclonal antibody.
  * At least 14 days after local palliative XRT (small port); At least 150 days must have elapsed if prior TBI, craniospinal XRT or if ≥ 50% radiation of pelvis; At least 42 days must have elapsed if other substantial bone marrow radiation.
  * No evidence of active graft vs. host disease and at least 84 days must have elapsed after transplant or stem cell infusion.
  * Patient must not have had prior exposure to gene vector delivery products within 3 months.
  * Patients may not have had prior SGT-53. Patient who have received prior topotecan, cyclophosphamide, or both are eligible.
* Adequate Bone Marrow Function:

  * Peripheral absolute neutrophil count (ANC) ≥ 1000/mm³.
  * Platelet count ≥ 100,000/mm³.
* Adequate Renal Function:

  * Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m² OR age/gender appropriate serum creatinine.
* Adequate Liver Function:

  * Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age.
  * SGPT (ALT) ≤ 110 U/L.
  * Serum albumin ≥ 2 g/dL.

Exclusion Criteria:

* Are pregnant or breast-feeding women.
* Concomitant medications:

  * Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible.
  * Patients who are currently receiving another investigational drug are not eligible.
  * Patients who are currently receiving other anti-cancer agents are not eligible.
  * Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial.
* Patients who have an uncontrolled infection are not eligible.
* Patients who have received a solid organ transplantation are not eligible.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-12; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) | 3-18 weeks
  The dose limiting toxicities of SGT-53 alone and in combination with topotecan and cyclophosphamide in pediatric patients with recurrent or refractory solid tumors will be assessed by any adverse events that are possibly, probably or definitely attributable to study drugs.
Recommended phase 2 dose (RP2D) | 3-18 weeks
  The recommended phase 2 dose of SGT-53 alone and in combination with topotecan and cyclophosphamide in pediatric patients with recurrent or refractory solid tumors will be assessed.

SECONDARY OUTCOMES:
Tolerability of systemic intravenous infusion (assessed by any adverse events related to infusion of study drugs according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.) | 3-18 weeks
  Tolerability of systemic intravenous infusion of SGT-53 alone and in combination with topotecan and cyclophosphamide will be assessed by any adverse events related to infusion of study drugs according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Anti-tumor activity (evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.) | 3-18 weeks
  Anti-tumor activity of SGT-53 alone and in combination with topotecan and cyclophosphamide will be evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.
Concentration of SGT-53 over time will be characterized by Cmax and clearance (Pharmacokinetic will be performed to evaluate the concentration of SGT-53 in patient's blood over time) | 3-18 weeks
  Pharmacokinetic will be performed to evaluate the concentration of SGT-53 in patient's blood over time

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Muscal, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States